CLINICAL TRIAL: NCT04874545
Title: Effect of Propfol Versus Sevoflurane on Auditory and Cognitive Function: A Compartive Study
Brief Title: Effect of Propfol Versus Sevoflurane on Auditory and Cognitive Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mona Hussein, Associate professor of Neurology, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: FMBSUREC/1206018/Abdelhamid
Record Dates: First submitted 2021-04-17; First posted 2021-05-05 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Cognitive Dysfunction; Auditory Dysfunction, Central
MeSH Terms: conditions — Cognitive Dysfunction; Auditory Diseases, Central | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol group (Experimental): Maintenance of anaesthesia will be done using Propofol total intravenous anesthesia (TIVA) 6-12 mg/ kg/h by syringe pump, 100 % O2.
  Interventions: Drug: Propofol
- sevoflurane group (Active Comparator): Maintenance of anaesthesia will be done using sevoflorane1.5-2%, 100 % O2.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Total intravenous inhalational anesthesia
  Other Names: Sevoflurane

SUMMARY:
Perioperative hearing loss is a rarely reported phenomenon. However, it occurs more frequently than most anaesthesiologists suspect. Perioperative hearing impairment is often subclinical and may go unnoticed unless audiometry is performed.

It can be conductive or sensorineural, unilateral or bilateral, and transient or permanent. Hearing loss has been reported following virtually every type of anaesthetic technique.

The hearing mechanism may be less susceptible to acoustic trauma during general anaaesthesia. But other mechanisms are capable of causing both conductive and sensorineural hearing losses (SNHL) in the perioperative period. The aetiologies include mechanical, traumatic, noise-induced, changes in cerebrospinal fluid (CSF) pressure, embolism, pharmacologic, and other miscellaneous causes.

Stress may influence central vestibular function in health and disease either directly through the actions of glucocorticoids (cortisol and corticosterone) on ion channels and neurotransmission in the brain, or indirectly through the effects of stress-related neuroactive substances (e.g., histamine, neurosteroids) on these structures.

The auditory brainstem response (ABR) provides a good estimate of the shape of the behavioral audiogram [and is thus an extremely useful tool for studying hearing sensitivity as well as the functionality of the auditory system.

An awareness of the potential for and the causes of hearing loss during anesthesia may permit the anesthesiologist to prevent or minimize the risk of significant hearing deficit. The suggestion that this risk be discussed in the preoperative period with patients who are at high risk for perioperative hearing loss may be good medical-legal advice. Better understanding of the incidence, causes, and prognoses for perioperative hearing loss is essential for the anesthesiologist.

Much Concern has been raised about the effects of anaesthetic drugs on cognition. Postoperative cognitive dysfunction may manifest as impairment in attention, memory, language or executive functions following surgery, and can persist for weeks, months, or more with varying severity. Such post-operative cognitive dysfunction can be quite mild and only diagnosed through psychometric assessment using specific neuropsychological tests.

AIM OF THE STUDY The aim of this work is to study the possible deleterious effect of propfol versus sevoflurane on auditory and cognitive function.

DETAILED DESCRIPTION:
Type and site of the study:

This study will be carried out at Beni-Suef university hospital, after approval by the department of Anaesthesiology, the local ethics and research committee and other involved departments, faculty of medicine, Beni-Suef University.

Date of the study:

The study will be performed starting from 1st of January 2021

Study design and population: This is a prospective randomized study that will be carried out on patients subjected to general anaesthesia.

Sampling Technique:

Patients will be randomly assigned into one of two equal groups Randomization will be carried out using a closed opaque envelope technique with the anesthetist will pick up a sealed envelope which contains a paper with the name of the group to which the patient will be randomized is written. Whichever the group written on the paper, the patient will be scheduled to it.

The patients will be subjected to the following:

* A routine preoperative check-up will be performed. Routine hematological and biochemical testing, along with electrocardiograms will be performed for patients. The procedure will be explained to the patients
* On arrival to the operating theatre, 18 G intravenous cannula will be inserted and IV crystalloid fluids will be infused, the monitor will be attached to the patients to take preoperative readings of heart rate, non-invasive arterial blood pressure, SpO2.
* The patients will be randomly divided to one of two groups:

Group 1:

* Induction of anesthesia will be done by injecting fentanyl 2 μg/kg, propofol1.5-2.5 mg/kg and atracurium 0.5 mg/kg for muscle relaxation. Laryngoscopy and endotracheal intubation will be performed using oral cuffed tube lubricated with lidocaine jelly 2 %.
* Maintenance of anaesthesia will be done using Propofol total intravenous anesthesia (TIVA) 6-12 mg/ kg/h by syringe pump, 100 % O2.

Group 2:

* Induction of anesthesia will be done by injecting fentanyl 2 μg/kg, propofol1.5-2.5 mg/kg and atracurium 0.5 mg/kg for muscle relaxation. Laryngoscopy and endotracheal intubation will be performed using oral cuffed tube lubricated with lidocaine jelly 2 %.
* Maintenance of anaesthesia will be done using sevoflorane1.5-2%, 100 % O2. The concentrations of propofol and sevoflorane will be adjusted according to patient's vital sign

Ventilation in both groups will be controlled artificially to maintain an end-tidal partial pressure of carbon dioxide of 33-35 mmHg.

At the end of surgery, neuromuscular blockade will be reversed with IV neostigmine 0.04mg/kg and atropine 0.02 mg/kg, the trachea will be extubated when the patient respond to commands, all patients will be transferred to PACU, where they receive oxygen via face mask 3-4 L/min and will be monitored.

The following parameters will be evaluated and recorded by senior anesthesiologist unaware of the study protocol:

1. Demographic data: age and sex
2. Operation type.
3. Duration of anesthesia
4. Hemodynamics of the patients: Mean arterial blood pressure and heart rate, SPO2, End tidal CO2: will be continuously monitored and recorded every 15 minutes

All included patients will be subjected to the following (preoperative and 1 week postoperative):

1) Cognitive assessment:

Cognitive functions for the patients will be assessed using the following psychometric tests:

1. Paired Associate Learning test (PALT) (9):

   * Aim: to assess auditory verbal memory. The test uses the concept of semantic cueing
   * Administration and scoring: In this test, the examiner says ten associated pairs in front of the candidate. These pairs contain 6 compatible semantically related pairs and 4 incompatible semantically unrelated pairs. After one minute, the candidate is given the first word of the pairs and is asked to recall the second word. The test is repeated three times. Each correct compatible pair takes a score 0.5, while each correct incompatible pair takes a score 1. The total score ranges from 0 to 21.
2. Paced Auditory Serial Addition Test (PASAT) ( 10):

   • Aim: Paced Auditory Serial Addition test is used for assessment of attention and auditory working memory

   • Administration and scoring: In this test, a series of 61 single digit numbers are spoken on an audiotape (or CD) at a rate of one every 3 seconds. The subject is asked to add each number to the one immediately preceding it and not to give a running total. The subject has to report the sum orally. Total score is the sum of correct responses and it ranges from 0 to 60.

2) Audiological assessment:

1. Audiological evaluation: tonal audiometry in the frequency range 0.25 - 8 kHz. Using orbiter 922 in a sound treated room with a TDH 39 earphones. Speech audiometry including speech reception threshold (SRT) using arabic spondee words, (11) and word discrimination score (WDS), using, arabic phonetically balanced (PB) words. (11) Immittancemetry: will be done using AD 629 Interacoustic, calibrated according to the ISO standard, using single-component, single-frequency tympanometry with a probe tone of 226 Hz. Testing of the acoustic reflex threshold, for ipsilateral and contralateral elicited reflexes, using pure tones at 500, 1000, 2000 and 4000 Hz.
2. Brainstem auditory evoked potentials (BAEPs): will be performed using (Interacoustic Eclipse ''EP25''). The reference electrodes will be placed on the right(A2) and left (Al) mastoids, the active is on the scalp at the vertex (Fz position of the 10-20 International System of EEG electrode placement) and the ground electrode is on the lower mid-frontal area (Fpz position). Ag/AgCl electrodes filled with conductive paste will be fixed to skin that will be abraded with a skin prepping gel. Electrode impedances will be less than 5 kΩ, and inter-electrode impedances will be less than 2 kΩ. The subject should be in relaxed state. Click is presented through TDH39 headphones. Click will be presented at a rate of 21.1 stimuli per second in rarefaction polarity at intensity of 80 dBHL. Averaged potentials to 1200 clicks will be obtained. Two recordings will be obtained to ensure the replicability of the waveforms. The latencies of waves I, III, V and interpeak latencies I-V, I- III, III-V (IPLs) will be studied with BAEPs.

'

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients who are candidate for elective extra cranial surgery.
* Male and female patients with age between 20-60 years

Exclusion Criteria:

* Patients with a conductive or sensorineural hearing loss
* Patients with a history of ear infection
* Patients with a history of ear trauma
* Patients using ototoxic or neurotoxic drugs
* Patients with sternocleidomastoid muscle pathology (traumatic injury or weakness) that interfere with audiological assessment
* Patient subjected to gross hemodynamic or ventilatory fluctuations during the operation
* Patient who developed postoperative shock or major bleeding
* Patient with a history of neurodegenerative disease, concomitant medical or metabolic illness known to affect cognition
* Allergy to any drug used in the study.
* Pregnancy.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Audiometry | 1 week
  A tool for assessment of auditory function
Paired associate learning test | 1 week
  A test for assessment of cognitive function
Paced Auditory Serial Addition Test | 1 week
  A test for assessment of cognitive function

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef University, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No